CLINICAL TRIAL: NCT03183817
Title: Person-centred Care at Distance for Persons With Chronic Heart Failure (CHF) and/or Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Person-centred Care at Distance
Acronym: PROTECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROTECT
Record Dates: First submitted 2017-06-07; First posted 2017-06-12 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure; Chronic Obstructive Pulmonary Disease
Keywords: Person-centred care
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Person-centred care at distance (Experimental): Person-centred care at distance through an eHealth platform, used both by professionals, patients and relatives
  Interventions: Behavioral: Person-centred care at distance
- Usual Care (No Intervention): Evidence-based care

INTERVENTIONS:
Behavioral: Person-centred care at distance — Person-centred care at distance through an eHealth platform
  Arms: Person-centred care at distance

SUMMARY:
The goal of the research project PROTECT is to translate the Person-Centred Care (PCC) principles into an eHealth (the use of information and communication technologies for health) context. A developed PCC eHealth platform will be used as a tool to identify patients´ resources to enhance coping and living with their chronic illness by means of a dialog and partnership with staff and relatives. The PCC eHealth platform will not replace, but instead be used as add on treatment to usual care (guideline directed care).

DETAILED DESCRIPTION:
A pilot study and collaboration between patients, relatives and professionals in the research program has clarified the need to develop a PCC eHealth platform. Previous research has shown that eHealth support, where the users are not involved in the process, has a low impact and has highlighted several limitations with respect to: patients' participation in the design process; its anchorage in the home and local environment and opportunities for communication rather than information. Therefore this study has a participatory design which assumes that all users (patients, relatives and health care professionals) are involved in the study design which facilitates implementation. An end-user perspective as a starting point increases the chances that users adapt a positive attitude towards the new system. Person-centred care combined with an eHealth support along the chain of health care showed a 4-fold chance of improved self-efficacy in combination with return to work or prior activity level after an event of acute coronary syndrome.

PCC can be delivered at distance and make health care more effective above and beyond usual care. Inclusion of the principles of PCC in an eHealth support for patients with chronic heart failure (CHF) and/or chronic obstructive pulmonary disease (COPD) will reduce the need for medical care (primary care and hospital admission) amongst these patients by improving self-management, self-efficacy and collaboration in the process of care.

The aim of this project is to implement and evaluate the PCC approach at distance to patients with CHF and/or COPD and their informal care givers to live better and cope more effectively with the disease burden associated with CHF and/or COPD. In the PCC approach, the aims, capabilities and needs of each patient, will be the starting point. Self-care strategies will be reinforced and empowered.

This study is a randomized, open, parallel group intervention study where patients are eligible when they are hospitalized due to worsening CHF and/or COPD. They will be asked before discharge about participation.

Patients admitted to hospital for worsening CHF and/or COPD will be recruited by the research nurses employed in this project from Emergency or on the ward once their condition has stabilized sufficiently.

Patients will be screened against inclusion and exclusion criteria for eligibility to participate in the study. Written informed consent will be obtained. Patients will be randomized into either the control or the intervention arm 1:1. The control group will receive usual care. The intervention group will receive usual care plus a PCC nurse-led intervention. Randomization will be done through computer generated lists and stored in sealed envelopes.

Patients listed in Närhälsan with a confirmed diagnosis of CHF and/or COPD will be screened and sent an informing letter about the study from the chief at each centre. Specially trained registered nurses (RNs) will then screen patients against study inclusion and exclusion criteria and by phone contact eligible patients and inform the patient about the aims of the study and ask if they are interested to participate. If the patient wants to participate a consent form is sent to the patient and then returned to the RN. Then the randomization procedure is performed which is based on a computer-generated list and the patient will be informed about the outcome by phone. Patients randomized to the intervention group will need a computer, smart phone or iPad to participate in the study. Patients who want will have the possibility to be provided an iPad for the duration of their participation in the programme.

Two dedicated full-time Registered Nurses (RN) follow the procedures closely. A monitor controls the protocol adherence. All case record forms, questionnaires and referrals will be constructed (for intervention and usual care groups).

Patients listed at a primary care centre in Närhälsan with CHF and/or COPD will be randomized to usual care (control) or PCC (intervention) after informed and written consent. Follow-up questionnaires on general self-efficacy, cardiac self-efficacy, quality of life, anxiety and depression will be sent out to all patients in both groups after 3,6,12 and 24 months after randomization.

Patients randomized to usual care will be managed by regular evidence-based treatment and care as outlined in treatment guidelines and followed as usual at their local primary care centre.

Patients will be called by a dedicated RN who has received special training in PCC communication at distance, the eHealth platform, CHF and COPD for an initial person-centred dialogue by phone. Based on the patient narrative patient´s goals, resources and needs are identified. The patient (sometimes maybe together with relatives) and the RN formulate a person-centred health plan. This plan is part of and will be up-loaded to the eHealth platform which also contains individual notes and information about CHF and COPD. The plan will be the point of departure for the forthcoming dialogue at distance via the eHealth platform that the patient and the RN will have during the study period (6 months).

The eHealth support contains headings that may inspire the patient to make notes on "a good day" respectively "a bad day". The health plan contain three parts; 1. "My goal is to feel or be able to do". 2. "To be able to reach my goal I will." 3."Support I need to reach my goal". In the communication during the study period between the RN and patient, the personal health plan is discussed and any needs of reformulating the goals may be discussed. The overall goal is to help the patient to identify their own capabilities/resources such as a strong will, social relations etc. and formulate goals that help them increase their self-efficacy and to cope with their condition in daily life.

The RN presents the eHealth support for communication (computer, iPad, smart phone) and they agree on how they will be in contact thereafter. The RN invites the patient and activates their account where he/she can login via an individual user name and formulate, comment, evaluate or develop the health plan. Access to the diary will be password protected. Different forms of symptom-ratings and comments can also be made. The RN can see the patient´s account and make comments. The patient can add or delete staff or private persons that have access to the account. The patient can also limit the access to the account. This makes it relatively simple to connect it to the health account (patient record through internet)

ELIGIBILITY:
Inclusion Criteria:

* National registration within the Västra Götaland Region (VGR)
* Men and women listed at a primary care centre in Närhälsan with a history of confirmed diagnosis of COPD and /or CHF
* Must understand written and spoken Swedish

Exclusion Criteria:

* Severe impairment that prevents patient from using the eHealth support
* No registered address
* Any severe disease with an expected survival < 12 months
* Cognitive impairment (SPMSQ score >6)
* Ongoing documented diagnosis of alcohol or drug abuse
* Other disease that can interfere with follow-up (e.g. severe depression, other severe mental illness)
* Patient participating in another conflicting randomized study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite score of changes in general self-efficacy | baseline, 3, 6, 12, 24 months
  The primary efficacy endpoint is a composite score of changes in general self-efficacy 18 based on the General Self-Efficacy Scale (GSE), hospitalization and death. The rationale for such an endpoint is the value of combining patient experience and clinical outcomes.
  A patient is classified as improved, deteriorated or unchanged:
  * A patient is classified as deteriorated if any of the following occurred:
    · at 6 months, self-efficacy has decreased by > 5 units (the minimal change of clinical significance) or has been admitted to hospital for unscheduled reasons or died.
  * A patient is classified as improved if:
    * self-efficacy has increased by > 5 units and has not been hospitalized.
  Those who have neither deteriorated nor improved are considered unchanged.

SECONDARY OUTCOMES:
Number of admissions | 3, 6, 12, 24 months
  Number of admissions
General self-efficacy scale | 3,6,12,24 months
  Questionnaire
Health care utilization | 3,6,12,24 months
  number of admissions and unscheduled outpatient visits due to unplanned visits to hospital and/or primary care centre due to symptoms of COPD and CHF
Incremental cost-utility ratios | 3,6,12, 24 months
  Incremental cost-utility ratios
Health-related quality of life (EQ-5D) | 3,6,12,24 months
  Questionnaire
Hospital anxiety and depression scale (HADS) | 3,6,12,24 months
  Questionnaire
Shortness of breath in heart failure (SOB-HF) | 3,6,12,24 months
  Questionnaire
COPD Assessment Test (CAT) | 3,6,12,24 months
  Questionnaire
The MRC breathlessness scale | 3,6,12,24 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Inger Ekman, Professor, Principal Investigator — Institute of health and care sciences, Centre for person-centred care (GPCC)
Locations (1):
- Primary health care, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barenfeld E, Ekman I, Cederberg M, Fors A, Ali L, Gyllensten H. Patient and healthcare professional engagement and time use within a randomised controlled trial: investigating intervention costs associated with remote person-centred care in Sweden. BMJ Open. 2025 Oct 9;15(10):e099034. doi: 10.1136/bmjopen-2025-099034. PMID 41067773
- [Derived] Harvey BP, Barenfeld E, Fors A, Ekman I, Swedberg K, Gyllensten H. Economic evaluation of a person-centred care intervention with a digital platform and structured telephone support for people with chronic heart failure and/or chronic obstructive pulmonary disease: results from a randomised controlled trial in Sweden. BMJ Open. 2025 Oct 9;15(10):e093083. doi: 10.1136/bmjopen-2024-093083. PMID 41067758
- [Derived] Ali L, Wallstrom S, Fors A, Barenfeld E, Fredholm E, Fu M, Goudarzi M, Gyllensten H, Lindstrom Kjellberg I, Swedberg K, Vanfleteren LEGW, Ekman I. Effects of Person-Centered Care Using a Digital Platform and Structured Telephone Support for People With Chronic Obstructive Pulmonary Disease and Chronic Heart Failure: Randomized Controlled Trial. J Med Internet Res. 2021 Dec 13;23(12):e26794. doi: 10.2196/26794. PMID 34898447
- [Derived] Poot CC, Meijer E, Kruis AL, Smidt N, Chavannes NH, Honkoop PJ. Integrated disease management interventions for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2021 Sep 8;9(9):CD009437. doi: 10.1002/14651858.CD009437.pub3. PMID 34495549
- [Derived] Ali L, Wallstrom S, Barenfeld E, Fors A, Fredholm E, Gyllensten H, Swedberg K, Ekman I. Person-centred care by a combined digital platform and structured telephone support for people with chronic obstructive pulmonary disease and/or chronic heart failure: study protocol for the PROTECT randomised controlled trial. BMJ Open. 2020 Jul 19;10(7):e036356. doi: 10.1136/bmjopen-2019-036356. PMID 32690519